CLINICAL TRIAL: NCT00949845
Title: An fMRI Study of Cytokine-Associated Depression and Social Pain
Brief Title: Cytokine-Associated Depression and Social Pain
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Naomi Eisenberger
Purpose: Basic Science
Other Study IDs: Endotoxin
Record Dates: First submitted 2009-07-29; First posted 2009-07-30 (Estimated); Last update posted 2009-07-30 (Estimated); Status verified 2009-07

CONDITIONS: Depression
Keywords: Effect of Inflammatory challenge on depressed mood; Effect of inflammatory challenge on social pain
MeSH Terms: conditions — Depression | interventions — Endotoxins

INTERVENTIONS:
Drug: Endotoxin

SUMMARY:
Recent research has demonstrated a relationship between depression and immune system activity, specifically proinflammatory cytokine activity. Although experimentally-induced immune activation leads to increases in depressed mood, the neural correlates associated with these changes have remained largely unexplored. Based on relationships between cytokine activity, depression, and heightened physical and social pain sensitivity, I propose to investigate the effect of proinflammatory cytokine activation on the neural correlates of socially painful experience that may contribute to depression. Our previous work has shown that the dorsal anterior cingulate cortex (dACC), typically associated with physical pain distress, also plays a role in the distressing feelings associated with social rejection or social loss. Moreover, recent pilot data has revealed that individuals with elevated levels of baseline proinflammatory cytokines report feeling more distressed and show more dACC activity during social rejection. To investigate the causal role that cytokines may play in the heightened social pain sensitivity that can contribute to depression, participants will be randomly assigned to receive either endotoxin (which increases proinflammatory cytokine activity) or placebo. Subsequently, participants will complete a neuroimaging study in which they will be rejected during an online ball-tossing game. We hypothesize that individuals exposed to endotoxin will report more social distress and depression following rejection and will show more dACC reactivity during rejection. The proposed study is the first to investigate the effect of systemic inflammation on neural reactivity related to social and affective processes that may increase the risk of depression.

ELIGIBILITY:
Inclusion Criteria:

* right-handed

Exclusion Criteria:

* 1) BMI greater than 30,
* 2) presence of physical health problems or medication use,
* 3) evidence of an Axis I psychiatric disorder based on the SCID assessment,
* 4) evidence of recreational drug use from a positive urine test,
* 5) positive pregnancy test, if female,
* 6) abnormalities on screening laboratory tests (blood cell count, liver function),
* 7) claustrophobia,
* 8) metal in body,
* 9) history of allergies, autoimmune, liver, or other severe chronic diseases,
* 10) current use of prescription medications,
* 11) nightshift work or time zone shifts (> 3hrs) within the previous 6 weeks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Dates: Start 2007-01

CONTACTS AND LOCATIONS:
Overall Officials: Naomi I Eisenberger, Ph.D., Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA General Clinical Research Center, Los Angeles, California, United States

REFERENCES:
- [Result] Eisenberger NI, Inagaki TK, Rameson LT, Mashal NM, Irwin MR. An fMRI study of cytokine-induced depressed mood and social pain: the role of sex differences. Neuroimage. 2009 Sep;47(3):881-90. doi: 10.1016/j.neuroimage.2009.04.040. Epub 2009 Apr 17. PMID 19376240
- [Derived] Eisenberger NI, Berkman ET, Inagaki TK, Rameson LT, Mashal NM, Irwin MR. Inflammation-induced anhedonia: endotoxin reduces ventral striatum responses to reward. Biol Psychiatry. 2010 Oct 15;68(8):748-54. doi: 10.1016/j.biopsych.2010.06.010. Epub 2010 Aug 16. PMID 20719303